CLINICAL TRIAL: NCT00278642
Title: High Dose Cyclophosphamide & ATG With Hematopoietic Stem Cell Support in Patients With Autoimmune Bullous Skin Disorders: A Phase I Trial
Brief Title: Hematopoietic Stem Cell Support in Patients With Autoimmune Bullous Skin Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor stopped the study because of lack of elligible participants
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD Derm.Auto2001
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stem cell transplantation (Experimental)
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation

SUMMARY:
Autoimmune Bullous Skin Disorders are believed to be due to immune cells, cells that normally protect the body and are now causing damage to the body. This study is designed to examine whether treating patients with high dose cyclophosphamide (a drug which reduces the function of the immune system) together with anti-thymocyte globulin (a protein that kills the immune cells that are thought to be causing your disease), followed by return of the previously collected special blood cells (stem cells) will result in improvement of this disease. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the intense chemotherapy is to destroy the cells in the immune system which may be causing this skin disease. The purpose of the stem cell infusion is to restore the body's blood production, which will be severely impaired by the high dose chemotherapy and anti-thymocyte globulin.

ELIGIBILITY:
Inclusion Criteria:

1. Less than chronologic age 60 years at the time of pre-transplant evaluation.
2. An established diagnosis of an autoimmune skin disorder that includes any of the following:

   1. pemphigus vulgaris
   2. pemphigus foliaceus

   Diagnosis of bullous skin lesions will be based on history and physical, skin biopsy (light microscopy and indirect fluorescence), indirect immunofluorescence titer, BP 180 and 230 titers, Desmolglein-3 and Desmoglein-1 antibody, and photograph.
3. Patients who failed corticosteroids (equivalent dosage of prednisone 0.5 mg/kg/day for more than 3 months), and at least two of the following: azathioprine, mycophenolate mofetil, gold, tetracycline (or minocycline), cyclosporin, methotrexate, gold, or plasmapheresis. Failure is defined as the inability to wean steroids to less than 0.5 mg/kg/day.
4. Potential candidates must have involvement of more than 10% of skin body surface area, involvement of one or more mucosal lesions, or recurrent infections requiring more than two hospitalizations in which the source of the infection was due to bullous skin disease.
5. All candidates must be evaluated by two dermatologists, Dr. Joan Guitart and Dr. Joaquin Brieva, who must concur that the patient has refractory disease that may, in their clinical judgement, be associated with a 5-10% mortality if not controlled.
6. A minimum of 2.0 x 106 CD34+ cells/kg after selection are necessary to proceed to transplant.

Exclusion Criteria:

1. Individuals less than 18 years of age.
2. Significant end organ damage such as:

   1. LVEF <40% or deterioration of LVEF during exercise test on MUGA or echocardiogram.
   2. Untreated life-threatening arrhythmia.
   3. Active ischemic heart disease or heart failure.
   4. DLCO <45% or FEV1/FEV < 50%.
   5. Serum creatinine > 2.5 mg/dl.
   6. Liver cirrhosis, transaminases >3x of normal limits or bilirubin >2.0 unless due to Gilberts disease.
3. HIV positive.
4. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
5. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
6. Positive pregnancy test, inability or unable to pursue effective means of birth control, or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
7. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
8. Inability to give informed consent.
9. Major hematological abnormalities such as platelet count less than 100,000/ul, or ANC less than 1000/ul.
10. Presence of infected skin lesions. All skin lesions should be free of suppurative exudate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2002-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percent surface area involved New skin or mucosal blister development Immune suppressive medication requirements Survival | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States